CLINICAL TRIAL: NCT00605241
Title: A Randomized, Double-bind, Placebo Controlled, Two-way Cross-over Study to Assess the Effects of a Single Dose of GSK598809, a Selective DRD3 Antagonist, in Modulating Nicotine Reward
Brief Title: A Study To Assess The Effects Of A Single Dose Of GSK598809 In Modulating Nicotine Reward
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DAN106593
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Substance Dependence
Keywords: pharmacodynamics,; pharmacokinetics,; tolerability,; Safety,; single dose,; placebo,; Nicotine reward; GSK598809
MeSH Terms: conditions — Substance-Related Disorders | interventions — GSK598809

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- GSK598809 (Other): Drug
  Interventions: Drug: GSK598809

INTERVENTIONS:
Drug: GSK598809 — Drug

SUMMARY:
GSK598809 is being developed as an innovative treatment for substance dependence and potentially other compulsive behavioral disorders. This study will asses the effects of a single dose of GSK598809 in modulating nicotine reward in 2 cohorts of otherwise healthy male volunteers who smoke. Each cohort of subjects will receive a single dose of placebo or GSK598809 in two dosing sessions binded crossover fashine. There will be a washout period of at least seven days between each session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male smokers aged 18-65 with a desire to quit smoking.
* Body weight greater than 50kg and BMI within range 19 - 29.9 kg/m2
* Healthy with no significant medical, psychiatric or laboratory evaluation abnormality.

Exclusion Criteria:

* Positive pre-study urine drug/breath alcohol screen: positive HIV 1/2, Hepatitis B or Hepatitis C test at screening.
* History of alcohol/drug abuse or dependence (other than nicotine) within 12 months of the study.
* History of psychiatric disorder or sensitivity to any of the study medications or components thereof or a history of drug or allergy that in the opinion of the physician responsible contraindicates their participation.
* History of cardiac or pulmonary disease/abnormalities.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-02-25 (Actual); Primary Completion 2009-03-20 (Actual); Study Completion 2009-03-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | through 24 hours

SECONDARY OUTCOMES:
Stroop test | through 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Mugnaini M, Iavarone L, Cavallini P, Griffante C, Oliosi B, Savoia C, Beaver J, Rabiner EA, Micheli F, Heidbreder C, Andorn A, Merlo Pich E, Bani M. Occupancy of brain dopamine D3 receptors and drug craving: a translational approach. Neuropsychopharmacology. 2013 Jan;38(2):302-12. doi: 10.1038/npp.2012.171. Epub 2012 Sep 12. PMID 22968817
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study DAN106593 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/DAN106593?search=study&search_terms=DAN106593#rs
- Available data/document: Individual Participant Data Set: DAN106593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: DAN106593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: DAN106593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: DAN106593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: DAN106593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: DAN106593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: DAN106593 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register